CLINICAL TRIAL: NCT06999928
Title: Pilot Implementation-Effectiveness Study of an Enhanced Mentor Mother Strategy
Brief Title: Enhanced Mentor Mother Strategy for Pregnant and Postpartum Women Living With HIV
Acronym: PIE-eMMs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James G. Carlucci, Assistant Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24102; K23HD109056 (NIH)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hiv; Transmission Vertical; Viremia; Adherence, Treatment; Stigmatization; Socioeconomic Adversity; Health Care Utilization; Health Care Acceptability; Peer Group; Mothers
Keywords: prevention of mother-to-child transmission; retention; implementation; mentor mothers; differentiated service delivery; maternal-child health; Kenya
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Viremia; Treatment Adherence and Compliance; Stereotyping; Financial Stress; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Pregnant and postpartum WLHIV will be screened for risk factors, then those with risk factors will received problem-focused MM support, while those without risk factors will receive less intensive MM support.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced Mentor Mother Strategy (Experimental): Participants will receive support from a Mentor Mother (MM) who delivers a risk-based, differentiated package of PMTCT services tailored to the needs of pregnant and postpartum women living with HIV (WLHIV). At each clinic visit, the MM will assess maternal and infant risk using a structured tool. Based on the result, the MM provides tailored support, such as counseling, navigation, linkage to resources, or increased follow-up. WLHIV without identified risks receive a streamlined support package. The strategy is integrated into routine antenatal and postnatal care at the study site.
  Interventions: Behavioral: Enhanced Mentor Mother Strategy

INTERVENTIONS:
Behavioral: Enhanced Mentor Mother Strategy — The enhanced Mentor Mother strategy introduces a structured approach to differentiated PMTCT support, led by trained peer counselors/Mentor Mothers (MM). Mentor Mothers will be trained on how to perform risk stratification, and they will use a standardized form to identify and document psychosocial and clinical risk factors. Based on these, MMs then deliver tailored interventions, including additional counseling, community outreach, and referrals. Fidelity assessments and a process of audit and feedback will be used to further refine the strategy, which builds on national differentiated service delivery guidelines and integrates into routine care without requiring added clinic staff.

SUMMARY:
Mentor Mothers (MMs) are peer supporters who help pregnant and postpartum women living with HIV (WLHIV) as they receive prevention of mother-to-child transmission of HIV (PMTCT) services in resource-limited settings like Kenya. Differentiated service delivery (DSD) is a care model that tailors services based on clients' needs, helping to improve both the quality and efficiency of care.

This hybrid implementation-effectiveness study will test whether an enhanced MM strategy that uses DSD can be successfully carried out and improve health outcomes for mothers and infants. The study will take place at Burnt Forest Sub-District Hospital (BFSDH) in Kenya.

Researchers will ask:

* Can the enhanced MM strategy be delivered as planned and accepted by patients and staff?
* Does the strategy improve clinical outcomes like keeping mothers in PMTCT care, achieving HIV viral suppression, completing infant HIV testing, and preventing HIV transmission to infants? Researchers will compare health outcomes before and after the strategy is introduced at BFSDH, and also compare outcomes at other similar clinics that continue with standard MM services.

Women who choose to participate will meet with a MM during their routine antenatal and postnatal clinic visits. They will be offered the enhanced MM support, but can choose to receive standard care if they prefer.

DETAILED DESCRIPTION:
This is a hybrid implementation-effectiveness study of an enhanced Mentor Mother (MM) strategy for delivering risk-based, differentiated prevention of mother-to-child transmission of HIV (PMTCT) services to pregnant and postpartum women living with HIV (WLHIV) and their infants. The study will be conducted at Burnt Forest Sub-District Hospital (BFSDH), an Academic Model Providing Access to Healthcare (AMPATH)-supported public health facility in Uasin Gishu County, Kenya.

Mentor Mothers (MMs) are peer advocates who support WLHIV in PMTCT programs, providing adherence counseling, psychosocial support, and retention assistance. Although MMs are a widely implemented, evidence-based intervention, current models generally do not differentiate services based on clients' individual risk profiles. The enhanced MM strategy evaluated in this study builds on the World Health Organization and Kenya Ministry of Health's recommendation for differentiated service delivery (DSD)-a patient-centered model that tailors services to individual needs.

This study will evaluate implementation outcomes (feasibility, acceptability, fidelity) while also gathering preliminary clinical effectiveness data of the enhanced MM strategy. The strategy includes structured, iterative risk stratification by MMs and PMTCT clinicians at each clinical encounter to identify clients at higher risk for poor PMTCT outcomes. Identified risk factors include HIV viremia, stigma and non-disclosure, and socioeconomic barriers. Based on the identified risk(s), MMs will deliver individualized, problem-focused support. WLHIV with no identifiable risk factors will receive a less-intensive service schedule aligned with national differentiated care guidelines.

Specific Aims:

* Aim 1: Use a mixed-methods approach to evaluate fidelity, feasibility, and acceptability of the enhanced MM strategy over a 15-month period. Data will include quantitative fidelity checklists, MM activity logs, chart audits, observation logs, and stakeholder focus group discussions.
* Aim 2: Assess preliminary effectiveness of the enhanced MM strategy on key maternal and infant outcomes using aggregate, routinely collected clinical data from AMPATH's medical record system. Outcomes include maternal retention in care, maternal HIV viral suppression, infant uptake of HIV diagnostic testing, and HIV vertical transmission. A within-site pre-post analysis will compare outcomes at BFSDH during the 12 months before and after implementation (excluding the first 3 months of roll out). A contemporaneous across-site analysis will compare outcomes at BFSDH (enhanced MM strategy) and three comparable clinics providing standard MM services during the same 12-month period.

The study is supported by the NIH through a K23 award (K23HD109056), and builds on extensive formative research, including qualitative interviews and human-centered design workshops with WLHIV, MMs, PMTCT clinicians, and policymakers. Pilot implementation is being guided by local stakeholders and is expected to inform the design of a future pragmatic trial. The enhanced MM strategy, if successful, may provide a scalable model for improving PMTCT outcomes in resource-constrained settings.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and postpartum women living with HIV (and their infants born during the study)
* ≥18 years of age
* Enrolled in PMTCT services at BFSDH
* Able to understand and provide informed consent in English or Kiswahili

Exclusion Criteria:

* Women who are not pregnant or postpartum
* <18 years of age
* Not enrolled in PMTCT services at BFSDH
* Unable to understand and provide informed consent in English or Kiswahili
* Cognitive impairment that would interfere with ability to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Fidelity: Proportion of enhanced Mentor Mother strategy tasks completed and services correctly assigned/delivered, as assessed by checklists, audits, and observations. | Fidelity to the enhanced MM strategy will be assessed throughout the 15-month implementation period, and a process of audit and feedback will be used to enhance fidelity and further refine the strategy.
  Fidelity is defined as the degree to which an intervention is implemented as intended. In this study, fidelity to the enhanced Mentor Mother (MM) strategy will be assessed using quantitative (checklists, audits) and qualitative (observations, logs) methods. A checklist of essential tasks will quantify adherence to MM workflows, calculated as the proportion of tasks completed out of those intended. Audits of clinical records, screening tools, and MM logs will assess accuracy of risk-based service delivery, calculated as the proportion of correctly assigned and delivered services. Direct observations will assess the quality of MM service delivery, and content logs will capture which MM components are delivered and how participants respond.
Acceptability: Participant ratings of acceptability of the enhanced Mentor Mother strategy, assessed by AIM scores, satisfaction surveys, and focus group discussions. | Acceptability of the enhanced MM strategy will be assessed at the end of the 15-month implementation period.
  Acceptability is the perception among implementation stakeholders that an intervention is agreeable or satisfactory. In this study, acceptability of the enhanced Mentor Mother (MM) strategy will be assessed using quantitative (questionnaires) and qualitative (focus group discussions) methods. The Acceptability of Intervention Measure (AIM) is a brief, validated questionnaire that will be administered to participants. A satisfaction survey will also be administered to identify parts of the strategy that cause frustration or other negative emotions and parts of the strategy that cause positive emotions. Results from AIM and satisfaction surveys will then be used to guide focus group discussions that will qualitatively assess perspectives about the acceptability of the enhanced MM strategy. Focus group discussions will be audio recorded, translated, and transcribed for thematic analysis.
Feasibility: Participant ratings of feasibility of the enhanced Mentor Mother strategy, assessed by FIM scores and focus group discussions. | Feasibility of the enhanced MM strategy will be assessed at the end of the 15-month implementation period.
  Feasibility is the extent to which an intervention can be successfully carried out within a given context. In this study, feasibility of the enhanced Mentor Mother (MM) strategy will be assessed using quantitative (questionnaires) and qualitative (focus group discussions) methods. The Feasibility of Intervention Measure (FIM) is a brief, validated questionnaire that will be administered to participants. Results from the FIM will then be used to guide focus group discussions that will qualitatively assess perspectives about the feasibility and readiness for scale-up of the enhanced MM strategy. Focus group discussions will be audio recorded, translated, and transcribed for thematic analysis.

SECONDARY OUTCOMES:
Proportion of mothers retained in care | Assessed at baseline (pre-implementation), 6-months (interim analysis), and at the end of the 15-month implementation period.
  Proportion of women living with HIV (WLHIV) enrolled in PMTCT services (those pregnant and ≤18 months postpartum) who were not lost to follow-up during the period of observation, excluding those who died or transferred out.
Proportion of mothers with HIV viral suppression | Assessed at baseline (pre-implementation), 6-months (interim analysis), and at the end of the 15-month implementation period.
  Proportion of WLHIV enrolled in PMTCT services who received antiretroviral therapy for at least 3 months, had at least one HIV viral load test, and never had a result >200 copies/ml during the period of observation.
Proportion of mothers who died | Assessed at baseline (pre-implementation), 6-months (interim analysis), and at the end of the 15-month implementation period.
  Proportion of WLHIV enrolled in PMTCT services who died during the period of observation.
Proportion of mothers who transferred out | Assessed at baseline (pre-implementation), 6-months (interim analysis), and at the end of the 15-month implementation period.
  Proportion of WLHIV enrolled in PMTCT services who transferred to another clinic during the period of observation.
Proportion of infants receiving HIV diagnostic testing | Assessed at baseline (pre-implementation), 6-months (interim analysis), and at the end of the 15-month implementation period.
  Proportion of infants with perinatal HIV exposure (those 0-18 months of age) who had their first HIV test performed by 10 weeks of age during the period of observation.
Proportion of infants infected with HIV (vertical transmission) | Assessed at baseline (pre-implementation), 6-months (interim analysis), and at the end of the 15-month implementation period.
  Proportion of infants with perinatal HIV exposure with any positive HIV DNA PCR test result between 0-18 months of age during the month period of observation.
Proportion of infants who died | Assessed at baseline (pre-implementation), 6-months (interim analysis), and at the end of the 15-month implementation period.
  Proportion of infants with perinatal HIV exposure who died during the period of observation.

CONTACTS AND LOCATIONS:
Locations (1):
- Burnt Forest Sub-District Hospital, Burnt Forest, Uasin Gishu County, Kenya

IPD SHARING:
Plan to Share IPD: No